CLINICAL TRIAL: NCT00161616
Title: A Prospective, Randomized, Controlled, Stratified Study of InductOs in Subjects With Open Diaphyseal Tibia Fractures Treated With Reamed Locked Intramedullary Nail Fixation
Brief Title: Study Evaluating InductOs in Diaphyseal Tibia Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 3100N8-400
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-07

CONDITIONS: Tibial Fractures
Keywords: Open Diaphyseal Tibia Fractures
MeSH Terms: conditions — Tibial Fractures | interventions — Bone Morphogenetic Protein 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): InductOs is rhBMP-2/ACS 1.5 mg/ml implanted once at the time of definitive fracture coverage +surgical fixation
  Interventions: Drug: InductOs
- B (Other): Standard of Care: Surgical fixation only
  Interventions: Drug: InductOs

INTERVENTIONS:
Drug: InductOs — InductOs is rhBMP-2/ACS 1.5 mg/ml implanted once at the time of definitive fracture coverage

SUMMARY:
Demonstrate a larger proportion of subjects with healed fractures among subjects treated with InductOs and reamed, locked intramedullary nailing compared to subjects treated with reamed, locked intramedullary nailing alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with acute open tibial shaft fractures (Gustilo Type I, II, IIIA, or IIIB) who require surgical management with reamed, statically locked intramedullary nail fixation and who are at low risk for amputation.
* Subjects should be at least 18 years of age, be skeletally mature, and be able to provide written informed consent.
* Initial fracture stabilization and wound debridement should occur within 1 day after injury and DFC should occur within 14 days after injury.

Exclusion Criteria:

* Planned treatment for the fracture should not include further procedures to promote fracture healing. After 16 weeks have elapsed since DFC, unanticipated procedures to promote fracture healing are permitted as clinically indicated.
* Presence of fracture distraction > 2 mm following definitive fracture fixation.
* Presence of purulent drainage from the fracture site or evidence of active osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, MedInfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Norway, Finland, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Study Chair — For UK/Great Britian, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com
Locations (24):
- Ghent, Belgium
- Turku, Finland
- France (2):
  - Créteil
  - Toulouse
- Germany (3):
  - Berlin
  - Mainz
  - Münster
- Italy (2):
  - Pavia
  - Roma
- Rotterdam, Netherlands
- Norway (2):
  - Bergen
  - Oslo
- Poland (4):
  - Bialystok
  - Lublin
  - Sosnowiec
  - Szczecin
- Bucharest, Romania
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Centurion
  - Durban
- Alcalá, Spain
- United Kingdom (2):
  - Bristol
  - Norwich

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from September 2003 to July 2007.
Pre-assignment Details: Assessment of the fractured limb was performed 24 hours before surgical fixation. Patients were stratified by severity of fracture (using Gustilo-Anderson Classification).
Groups:
- rhBMP-2/ACS: InductOs (dibotermin alfa) contains 12 mg of recombinant human bone morphogenetic protein-2 (rhBMP-2) in the form of a 1.5 mg/ml solution on an absorbable collagen sponge (ACS) implanted once at the time of definitive fracture coverage + surgical fixation
- Standard of Care: Standard of Care: Surgical fixation only
Period: Overall Study
Arm/Group | rhBMP-2/ACS | Standard of Care
Started | 139 | 138
Completed | 113 | 119
Not Completed | 26 | 19
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 17 | 13
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rhBMP-2/ACS | Standard of Care | Total
Number analyzed (Participants) | 139 | 138 | 277
Age Continuous [Mean (Standard Deviation); unit: years] | 39.48 (15.40) | 37.54 (14.87) | 38.52 (15.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 113 | 111 | 224

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Healed Fractures
Description: Patients categorized by investigator as healed, not healed, no outcome (using pre-specified criteria). Healed: no tenderness at fracture site or pain with weight bearing, presence of bridging callus or disappearance of fracture lines, no hardware failure, no secondary intervention to promote fracture healing. Not healed: diagnosis of delayed union or nonunion, hardware failure, secondary intervention procedure for fracture healing recommended or performed, or conduct of procedure that may interfere with fracture healing. No outcome: subjects who did not achieve either healed or not healed.
Time Frame: 13 and 20 weeks
Population: All patients randomized were analyzed.
Measure: Number; unit: patients
Arm/Group | rhBMP-2/ACS | Standard of Care
Number analyzed (Participants) | 139 | 138
patients
  Week 13 Healed | 83 | 66
  Week 13 Not healed | 8 | 13
  Week 13 No outcome | 48 | 59
  Week 20 Healed | 95 | 92
  Week 20 Not healed | 29 | 28
  Week 20 No outcome | 15 | 18
Statistical Analysis 1: Comparison: rhBMP-2/ACS vs Standard of Care; Comparison of Healed vs Not healed/No outcome for week 13; Test type: Superiority or Other; p = 0.0541, Fisher Exact
Statistical Analysis 2: Comparison: rhBMP-2/ACS vs Standard of Care; Comparison of Healed vs Not healed/No outcome for week 20; Test type: Superiority or Other; p = 0.7983, Fisher Exact

2. Secondary Outcome: Number of Patients Achieving Combined Clinical and Radiographic Endpoint (CCRE)
Description: Patients categorized as Success or Failure of CCRE. Success defined as a fracture judged to be both clinically healed by clinical investigator, "healed" (see primary outcome), and radiographically united by independent, blinded radiology panel, "united." Patients deemed "not healed" or "not united" were assessed as failures.
Time Frame: 1 year
Population: All patients randomized were analyzed.
Measure: Number; unit: patients
Arm/Group | rhBMP-2/ACS | Standard of Care
Number analyzed (Participants) | 139 | 138
patients
  Success | 98 | 96
  Failure | 41 | 42
Statistical Analysis 1: Comparison: rhBMP-2/ACS vs Standard of Care; Test type: Superiority or Other; p = 0.8961, Fisher Exact

ADVERSE EVENTS:
Arm/Group | rhBMP-2/ACS | Standard of Care
Serious Adverse Events (participants affected / at risk) | 31 | 25
Other Adverse Events (participants affected / at risk) | 127 | 123
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | rhBMP-2/ACS | Standard of Care
Abcess (General disorders) | 0/139 | 1/138
Accidental injury (General disorders) | 2/139 | 4/138
Cellulitis (General disorders) | 1/139 | 0/138
Chest pain (General disorders) | 1/139 | 0/138
Fever (General disorders) | 1/139 | 0/138
Hardware failure (General disorders) | 0/139 | 2/138
Infection (General disorders) | 15/139 | 7/138
Pain (General disorders) | 7/139 | 2/138
Peritonitis (General disorders) | 1/139 | 0/138
Withdrawal syndrome (General disorders) | 0/139 | 1/138
Deep vein thrombosis (Vascular disorders) | 0/139 | 1/138
Embolus (Vascular disorders) | 1/139 | 0/138
Pulmonary embolus (Vascular disorders) | 1/139 | 0/138
Shock (Cardiac disorders) | 0/139 | 1/138
Intestinal obstruction (Gastrointestinal disorders) | 2/139 | 0/138
Anemia (Blood and lymphatic system disorders) | 0/139 | 1/138
Healing abnormal (Metabolism and nutrition disorders) | 0/139 | 1/138
Healing abnormal: bleeding at wound site (Metabolism and nutrition disorders) | 0/139 | 1/138
Healing abnormal: delayed wound healing (Metabolism and nutrition disorders) | 0/139 | 1/138
Healing abnormal: drainage, oozing, discharge (Metabolism and nutrition disorders) | 1/139 | 1/138
Healing abnormal: superficial wound breakdown (Metabolism and nutrition disorders) | 0/139 | 1/138
Hyperglycemia (Metabolism and nutrition disorders) | 0/139 | 1/138
Hypocalcemia (Metabolism and nutrition disorders) | 0/139 | 1/138
Peripheral edema (Metabolism and nutrition disorders) | 1/139 | 1/138
SGPT increased (Metabolism and nutrition disorders) | 0/139 | 1/138
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/139 | 0/138
Arthritis (Musculoskeletal and connective tissue disorders) | 0/139 | 1/138
Bone disorder (Musculoskeletal and connective tissue disorders) | 0/139 | 1/138
Bone fracture spontaneous (Musculoskeletal and connective tissue disorders) | 1/139 | 0/138
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 2/139 | 4/138
Fracture malalignment (Musculoskeletal and connective tissue disorders) | 2/139 | 3/138
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0/139 | 4/138
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1/139 | 0/138
Delirium (Nervous system disorders) | 0/139 | 1/138
Dizziness (Nervous system disorders) | 0/139 | 1/138
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/139 | 0/138
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/139 | 0/138
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1/139 | 0/138
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0/139 | 1/138
Skin necrosis (Skin and subcutaneous tissue disorders) | 0/139 | 1/138
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/139 | 0/138
Prostatic carcinoma (Reproductive system and breast disorders) | 1/139 | 0/138
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | rhBMP-2/ACS | Standard of Care
Fever (General disorders) | 8/139 | 8/138
Hardware failure (General disorders) | 24/139 | 20/138
Infection (General disorders) | 28/139 | 17/138
Lab test abnormal (General disorders) | 13/139 | 10/138
Pain (General disorders) | 88/139 | 84/138
Anemia (Blood and lymphatic system disorders) | 33/139 | 23/138
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 13/139 | 13/138
Amylase increased (Metabolism and nutrition disorders) | 10/139 | 7/138
Hyperglycemia (Metabolism and nutrition disorders) | 10/139 | 10/138
Hypocalcemia (Metabolism and nutrition disorders) | 11/139 | 12/138
Hypokalemia (Metabolism and nutrition disorders) | 6/139 | 8/138
Hypophosphatemia (Metabolism and nutrition disorders) | 6/139 | 15/138
Lactic dehydrogenase increased (Metabolism and nutrition disorders) | 27/139 | 26/138
Peripheral edema (General disorders) | 37/139 | 40/138
SGOT increased (Metabolism and nutrition disorders) | 24/139 | 23/138
SGPT increased (Metabolism and nutrition disorders) | 16/139 | 13/138
Arthralgia (Musculoskeletal and connective tissue disorders) | 16/139 | 7/138
Fractured delayed union (Musculoskeletal and connective tissue disorders) | 10/139 | 15/138
Post operative heterotopic calcification (Musculoskeletal and connective tissue disorders) | 13/139 | 8/138
Hypesthesia (General disorders) | 11/139 | 6/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.